CLINICAL TRIAL: NCT00170391
Title: Does CBT for Insomnia Improve the PSG Sleep of Patients Treated in Primary Care?
Brief Title: Do People With Insomnia Sleep Better After Psychological Treatment?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Organization: NHS Greater Clyde and Glasgow (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02CP08; 32966/1
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2002-10

CONDITIONS: Insomnia
Keywords: Insomnia; Sleep; PSG; Behavioural treatment
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

INTERVENTIONS:
Behavioral: Quarter of an Hour rule

SUMMARY:
The principal aim of the study is to evaluate if CBT for insomnia is associated with improvement in the PSG sleep of patients treated in primary care. Furthermore,the relationship between subjectively-assessed sleep and PSG sleep are investigated(at pre-treatment, at post-treatment, in relation to treatment change.

ELIGIBILITY:
Inclusion Criteria:

Meets clinical/RDC criteria for primary insomnia Healthy Adult (18+ years)

Exclusion Criteria:

Evidence of sleep disorders other than insomnia Use of sleeping pills Major Psychopathologies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2002-10; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Colin A Espie, PhD, Principal Investigator — University of Glasgow
Locations (1):
- Sackler Foundation of Psychobiological Research, Glasgow, Lanarkshire, United Kingdom